CLINICAL TRIAL: NCT00645892
Title: Extension Study of Two Dosing Schedules of Adalimumab in Subjects With Moderate to Severe Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Beverly Paperiello / Director, Clinical Program Management, Abbott
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M03-596
Record Dates: First submitted 2008-03-25; First posted 2008-03-28 (Estimated); Last update posted 2008-03-28 (Estimated); Status verified 2008-03

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: adalimumab
- B (Placebo Comparator)
  Interventions: Drug: placebo for adalimumab

INTERVENTIONS:
Drug: adalimumab — OL 80 mg at Weeks 0 and 1, 40 mg weekly Week 2 - Week 11, blinded 40 mg eow through Week 24
  Other Names: ABT-D2E7; Humira
  Arms: A
Drug: placebo for adalimumab — OL 80 mg at Weeks 0 and 1, 40 mg weekly Week 2 - Week 11, blinded placebo eow through Week 24
  Other Names: placebo
  Arms: B

SUMMARY:
Extension Study of Two Dosing Schedules of Adalimumab in Subjects with Moderate to Severe Chronic Plaque Psoriasis

ELIGIBILITY:
Inclusion Criteria:

* Subject participated and relapsed in prior PS study

Exclusion Criteria:

* Subject has other active skin diseases
* Multiple concomitant therapy restrictions and/or washouts (topicals, UV, other systemic PS therapies)
* Poorly controlled medical conditions
* History of neurologic symptoms suggestive of central nervous system (CNS) demyelinating disease.
* History of cancer or lymphoproliferative disease
* History of active TB or listeriosis, or persistent chronic or active infections
* Known to have immune deficiency or is immunocompromised
* Clinically significant abnormal laboratory test results
* Erythrodermic psoriasis or generalized pustular psoriasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2003-11; Primary Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Psoriasis Area and Severity Index | Week 12
Adverse Events | Throughout Study Participation

SECONDARY OUTCOMES:
Psoriasis Area and Severity Index | Week 12, Week 24
Physician's Global Assessment | Week 12, Week 24